CLINICAL TRIAL: NCT01590823
Title: Phase 1 Study of the Pharmacokinetics and Pharmacodynamics of Oral Dabigatran Etexilate in Hemodialysis Patients
Brief Title: An Evaluation of the Pharmacokinetics and Pharmacodynamics of Oral Dabigatran Etexilate in Hemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Capital Health, Canada (Other); Dalhousie University (Other); Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dabigatran Hemodialysis 2012
Record Dates: First submitted 2012-04-20; First posted 2012-05-03 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-04

CONDITIONS: Blood Coagulation Disorders
Keywords: pharmacokinetics
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dabigatran etexilate 110 mg (Other): Single dose of Dabigatran etexilate 110 mg po
  Interventions: Drug: Dabigatran Etexilate 110 mg

INTERVENTIONS:
Drug: Dabigatran Etexilate 110 mg — All participants will receive a single dosage of dabigatran etexilate 110 mg at the start of their 4 hour dialysis session. Blood sampling will be conducted during and up to 48 hours after participant's dialysis session.
  Other Names: Dabigatran Etexilate 110 mg (Pradax)

SUMMARY:
Patients with end stage renal disease carry a high risk for atrial fibrillation (AF) and require oral anticoagulant therapy for prevention of stroke. Often, the oral anticoagulant, warfarin sodium, is prescribed. Managing dialysis patients on warfarin can be fraught will difficulties given the multitude of drug and food interactions, need for frequent coagulation monitoring and dosage adjustment, and concern that warfarin enhances vascular calcification in dialysis patients. Recently, dabigatran etexilate, a direct oral thrombin inhibitor, has been approved for use in AF patients with normal renal function. Since many drugs are eliminated by the kidneys and removed from the plasma during dialysis, it is important to determine proper drug dosing in hemodialysis patients through evaluating pharmacokinetics.

DETAILED DESCRIPTION:
The frequency of atrial fibrillation (AF) is 10- to 20- fold higher in patients with end stage renal disease (ESRD) compared to the general population (1-5). Conditions contributing to the risk of stroke in AF are highly prevalent in ESRD patients undergoing dialysis (6). A large number of trials have shown the usefulness of oral anticoagulation with warfarin sodium for primary and secondary prevention of stroke in patients with AF (7). Despite that the majority of these trials excluded patients with ESRD, warfarin sodium is commonly prescribed in dialysis patients with AF for prevention of stroke (8). Managing dialysis patients on wafarin sodium is challenging given the plethora of drug and food interactions, need for frequent coagulation monitoring and dose adjustment and lack of large randomized clinical trails assessing the benefit of stroke prevention versus risk of hemorrhage in this population (8,9). Additionally, recent concern regarding the association between vascular calcification enhanced by warfarin sodium in dialysis patients highlights the need for alternative oral anticoagulant therapy (10,11).

A new oral anticoagulant, dabigatran etexilate, which is a direct thrombin inhibitor, has been approved for prevention of stroke in patients with AF and prevention of venous thromboembolic events (VTE) in patients who have undergone elective total hip and knee replacement surgeries(12-15). Other indications under investigation include the treatment of VTE (16) and the treatment of thromboembolic complications following acute coronary syndromes (17).

Dabigatran etexilate is an orally administered prodrug, which is rapidly absorbed and converted to its active form, dabigatran. Dabigatran specifically and reversibly inhibits thrombin which is a key enzyme required in the coagulation pathway. Dabigatran etexilate posses beneficial properties including: a fixed oral dosage regimen, predictable pharmacokinetic profile, strong association between plasma drug concentration and anticoagulation response, low potential for drug interactions and lack of need for routine coagulation monitoring (18-24). As such, dabigatran etexilate represents a possible improved alternative to warfarin for anticoagulation in dialysis patients with AF.

Dabigatran etexilate has been developed using a fixed dosage regimen of 150 mg twice daily in AF patients with normal renal function for prevention of stroke (12). Limited information regarding dosing dabigatran etexilate in patients with renal impairment or ESRD exists as these patients were excluded from all phase III trials. Despite this, a recent small study investigated the pharmacokinetics of a single oral dose of dabigatran etexilate 150 mg in healthy patients and in patients with mild to severe renal impairment (creatinine clearance >50 to ≤80 , >30 to ≤50 and <30 mL/min) and dabigatran etexilate 50 mg in patients with ESRD requiring maintenance hemodialysis (25).

Systemic exposure to dabigatran and corresponding coagulation response was increased by renal impairment and correlated with the severity of renal dysfunction suggesting that a reduced dose and or extended dose interval may be necessary in patients with mild to severe renal impairment. In the six patients that were studied, hemodialysis removed on average 62% and 68% of the dabigatran entering the dialyzer indicating that hemodialysis can compensate for the impaired dabigatran renal elimination that occurs in ESRD. Unfortunately, a meaningful correlation between dabigatran plasma concentrations and anticoagulation activity could not be determined as the hemodialysis patients were on unfractionated heparin to prevent clotting in their dialysis circuit. Furthermore, the necessity of a post-dialysis dose to maintain dabigatran levels in the therapeutic range was not investigated.

Herein, we propose a pilot study to examine the single dose pharmacokinetics and pharmacodynamics of dabigatran etexilate in hemodialysis patients who are receiving normal saline flushes for prevention of extracorporeal circuit clotting. The specific objective is to establish baseline correlation between plasma dabigatran concentrations versus anticoagulation activity over time. Our long-term objective is to develop an evidence-based recommendation for dabigatran dosing in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years receiving hemodialysis at the Capital District Health Authority Renal Program who are receiving or who are good candidates for normal saline flushes for prevention of extracorporeal circuit clotting will be eligible for this study.

Exclusion Criteria:

* Of those fulfilling the inclusion criterion, the following will be excluding characteristics:

  1. know bleeding diathesis;
  2. geographic inaccessibility for follow-up of timed blood sampling;
  3. use of any anticoagulant drugs that might influence results within 48 hours of the study;
  4. history of allergy/hypersensitivity (including drug allergy) deemed relevant to the trial by the investigators;
  5. recent or planned diagnostic or therapeutic procedures with potential for bleeding within 14 days before or after drug administration;
  6. history of familial bleeding disorder;
  7. history of relevant orthostatic hypotension, fainting spells or blackouts;
  8. disease of the central nervous system (such as epilepsy);
  9. chronic or relevant acute infection; and
  10. use of medication known to potentially increase or decrease dabigtran exposure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics following a single dose of dabigatran etexilate in hemodialysis patients. | 0,0.5,1,2,3,4,12,24, and 48 hours post dose following single dabigatran dose
  Dabigatran plasma concentration following a single dose of dabigatran etexilate in hemodialysis patients

SECONDARY OUTCOMES:
Fraction of dabigatran in the blood removed by dialysis. | 0,1,2,3 and 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: jo-anne wilsoon, PharmD, Principal Investigator — CDHA Renal Program
Locations (1):
- Capital Health District Authority, Department of Medicine, Division of Nephrology, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Wilson JA, Goralski KB, Soroka SD, Morrison M, Mossop P, Sleno L, Wang Y, Anderson DR. An evaluation of oral dabigatran etexilate pharmacokinetics and pharmacodynamics in hemodialysis. J Clin Pharmacol. 2014 Aug;54(8):901-9. doi: 10.1002/jcph.335. Epub 2014 May 28. PMID 24846496